CLINICAL TRIAL: NCT04539756
Title: Does an Online Two-week Positive Psychological Intervention Improve Positive Affect in Young Adults?
Brief Title: Writing Activities and Emotions
Acronym: eWrite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Caitlin M. DuPont, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY20060287
Record Dates: First submitted 2020-08-31; First posted 2020-09-07 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: Positive Psychological Intervention; Wellbeing; Optimism

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel study, such that participants are assigned to either an active control group or intervention group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active control condition (Active Comparator): Participants in the active control condition will receive the same number of text message reminders and will complete the same number of writing activities as the intervention group. The writing activity for the active control condition will ask them to list their activities for that day.
  Interventions: Behavioral: Active control condition
- Positive psychological intervention (Experimental): Participants will be asked to complete writing activities every other day. They will choose which activity they would like to complete each day, from a menu of six different activities. Each activity is a different positive psychology exercise.
  Interventions: Behavioral: positive psychological intervention

INTERVENTIONS:
Behavioral: positive psychological intervention — Participants will be asked to complete writing activities every other day. They will choose which activity they would like to complete each day, from a menu of six different activities. Each activity is a different positive psychology exercise.
  Other Names: Positive psychology exercises
  Arms: Positive psychological intervention
Behavioral: Active control condition — Participants will be asked to complete the same writing activity each day, which will ask them to list their daily activities. Participants will be encouraged to process their daily activities superficially by the receiving the following instructions: (1) list each activity in brief, incomplete sentences, (2) document only facts about performing the activities, and (3) to not provide any information about emotional responses to performing the activities. By following these instructions, participants are presumably deriving less meaning from their activities, which may minimize gains in positive affect in the active control condition
  Other Names: placebo
  Arms: Active control condition

SUMMARY:
The current study aims to test whether an online two-week positive psychological intervention can increase positive affect in college students. Participants will be recruited from the University of Pittsburgh undergraduate subject pool. Students will be ineligible if they are under the age of 18; currently prescribed medications for cardiac arrythmias; have a history of heart surgery, heart attack, or stroke; are currently pregnant; or currently have symptoms consistent with COVID-19. This study includes an active control arm and an intervention arm. Both arms will be required to complete writing activities every other day for two weeks. Participants in the control arm will list their daily activities, while participants in the intervention arm will complete various positive psychology activities. Questionnaires assessing mood, emotional well-being, social functioning and a few health behaviors will be administered pre- and post-intervention. The investigators aim to recruit 250 undergraduate students with the hope that at least 50 participants per group will complete the entire study.

ELIGIBILITY:
Inclusion Criteria:

* Must be an undergraduate student at the University of Pittsburgh that is currently taking Introduction to Psychology.
* Must be at least 18 years old
* Not currently prescribed medications for cardiac arrythmias
* Report no history of heart surgery, heart attack, or stroke
* Not currently pregnant
* Must deny having current symptoms consistent with COVID-19.

Exclusion Criteria:

* If the participant does not meet the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in positive affect at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  Positive and Negative Affective Schedule (20-item). The possible range for this questionnaire is from 5 - 50. Baseline values will be subtracted from post-intervention values and a higher score on this measure represents a better outcome.
Change from baseline in positive affect at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  Positive Emotional Style Questionnaire. The possible range for this questionnaire is from 0 - 36. Baseline values will be subtracted from post-intervention values and a higher score on this measure represents a better outcome.

SECONDARY OUTCOMES:
Change from baseline in optimism at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  Life Orientation Test-Revised. The possible range for this questionnaire is from 6 - 30. Baseline values will be subtracted from post-intervention values and a higher score on this measure represents a better outcome.
Change from baseline in life satisfaction at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  PROMIS - General Life Satisfaction. The possible range for this questionnaire is from 10 - 70. Baseline values will be subtracted from post-intervention values and a higher score on this measure represents a better outcome.
Change from baseline in psychological well-being at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  Psychological Well-Being Scale. The possible range for this questionnaire is from 42 - 294. Baseline values will be subtracted from post-intervention values and a higher score on this measure represents a better outcome.
Change from baseline in perceived stress at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  Perceived Stress Scale. The possible range for this questionnaire is from 0 - 40. Baseline values will be subtracted from post-intervention values and a higher score on this measure represents a worse outcome.
Change from baseline in perceived social support at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  ISEL (12-item). The possible range for this questionnaire is from 12 - 48. Baseline values will be subtracted from post-intervention values and a higher score on this measure represents a better outcome.
Change from baseline in loneliness at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  UCLA Loneliness Scale (8-item). The possible range for this questionnaire is from 0 - 24. Baseline values will be subtracted from post-intervention values and a higher score on this measure represents a worse outcome.
Change from baseline in depressive symptoms at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  PROMIS - Emotional Distress - Depression - Short Form. The possible range for this questionnaire is from 8 - 40. Baseline values will be subtracted from post-intervention values and a higher score on this measure represents a worse outcome.
Change from baseline in anxiety symptoms at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  PROMIS - Emotional Distress - Anxiety - Short Form. The possible range for this questionnaire is from 7 - 35. Baseline values will be subtracted from post-intervention values and a higher score on this measure represents a worse outcome.
Change from baseline in light physical activity (in general) at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  1-items asking participants to report minutes of light physical activity that they perform 'in general.' Baseline values will be subtracted from post-intervention values and a higher number on this measure represents a better outcome.
Change from baseline in moderate physical activity (in general) at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  1-item asking participants to report minutes of moderate to vigorous physical activity that they perform 'in general.' Baseline values will be subtracted from post-intervention values and a higher number on this measure represents a better outcome.
Change from baseline in sleep quality (in general) at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  1-item asking participants to report their overall sleep quality in general. Sleep quality was assessed on a Likert scale from Very bad (0) to Very good (5). Higher scores reflect a better outcome.
Change from baseline in sleep quantity (in general) at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  1-items asking participants to report how long they typically sleep each night.
Change from baseline in negative affect at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  Positive and Negative Affective Schedule. The possible range for this questionnaire is from 5 - 50. Baseline values will be subtracted from post-intervention values and a higher score on this measure represents a better outcome.
Change from baseline in negative affect at 1 week post-intervention | Assessed twice, once before the intervention and a second time within one week of completing the intervention.
  Negative Emotional Style Questionnaires. The possible range for this questionnaire is from 0 - 36. Baseline values will be subtracted from post-intervention values and a higher score on this measure represents a worse outcome.

OTHER OUTCOMES:
Loneliness | Assessed every other day, after participants complete each activity for up to 2 weeks.
  Participants will be asked to rate how much they agree with the following statement on a visual analogue scale from "Not at all accurate (0)" to "Extremely Accurate (100)". The statements states: Today I feel lonely or isolated. Higher scores reflect worse outcomes.
Connectedness | Assessed every other day, after participants complete each activity for up to 2 weeks.
  Participants will be asked to rate how much they agree with the following statement on a visual analogue scale from "Not at all accurate (0)" to "Extremely Accurate (100)". The statements states: Today I feel connected to others. Higher scores reflect better outcomes.
Stress | Assessed every other day, after participants complete each activity for up to 2 weeks.
  Participants will be asked to rate how much they agree with the following statements on a visual analogue scale from "Not at all accurate (0)" to "Extremely Accurate (100)". Stress will be assessed by the one-item statement: 'Today I feel stressed.' Higher scores reflect worse outcomes.
School-specific stress | Assessed every other day, after participants complete each activity for up to 2 weeks.
  Participants will be asked to rate how much they agree with the following statements on a visual analogue scale from "Not at all accurate (0)" to "Extremely Accurate (100)". School stress will be assessed by the one-item statement: 'Today I feel nervous or overwhelmed about school.' Higher scores reflect worse outcomes.
Light physical activity (today) | Assessed every other day, after participants complete each activity for up to 2 weeks.
  Participants will self-report minutes of light physical activity that they completed that day. Larger numbers reflect better outcomes.
Moderate to vigorous physical activity (today) | Assessed every other day, after participants complete each activity for up to 2 weeks.
  Participants will self-report minutes of moderate to vigorous physical activity that they completed that day. Larger numbers reflect better outcomes.
Sleep quantity (today) | Assessed every other day, after participants complete each activity for up to 2 weeks.
  1-items asking participants to report how long they slept the night before.
Sleep quality (today) | Assessed every other day, after participants complete each activity for up to 2 weeks.
  Sleep quality was assessed on a 1-item Likert scale asking participants to rate their subjective sleep quality from Very bad (0) to Very good (5). Larger numbers represent better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin M DuPont, MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
I do not plan on sharing any of the individual participant data with other researchers.